CLINICAL TRIAL: NCT06931145
Title: A Real-world Study of Benmelstobart, Anlotinib and Chemotherapy Regimen as First-line Treatment for Extensive-stage Small-cell Lung Cancer
Brief Title: Benmelstobart, Anlotinib and Chemotherapy as First-line Treatment for Extensive-stage Small-cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Wang mengzhao, chief physician, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K7820
Record Dates: First submitted 2025-04-09; First posted 2025-04-17 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Extensive-stage Small Cell Lung Cancer
Keywords: small cell lung cancer; benmelstobart; anlotinib
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — anlotinib; Carboplatin; Cisplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Benmelstobart in combination with anlotinib and chemotherapy (Experimental): Patients who met the enrollment criteria were first treated with benmelstobart in combination with anlotinib and carboplatin/cisplatin and etoposide for 4 cycles, and for non-progressing patients were evaluated by the investigator to receive maintenance therapy with benmelstobart in combination with anlotinib, which was continued until clinical benefit was lost or toxicity was intolerable or efficacy was evaluated to be PD, or continuation of the medication was deemed unsuitable by the investigator.
  Interventions: Drug: Benmelstobart; Drug: Anlotinib; Drug: Carboplatin or cisplatin; Drug: Etoposide

INTERVENTIONS:
Drug: Benmelstobart — Benmelstobart injection, 1200 mg/dose, given once every 21 days, intravenously.
Drug: Anlotinib — Anlotinib hydrochloride capsules, 8 mg/dose, administered orally for 2 consecutive weeks and stopped for 1 week.
  During the course of the study, subjects may be adjusted upward to a dose of 12 mg if well tolerated, as determined by the investigator, and the dose of anlotinib hydrochloride may be adjusted downward during the course of the study due to drug-related adverse events.
Drug: Carboplatin or cisplatin — Carboplatin for injection, administered on day 1, AUC 5 mg/mL/min, intravenously (maximal dose used is 750 mg); or cisplatin administered on day 1, 75-80mg/m2, IV.
Drug: Etoposide — Etoposide injection, 100mg/m2 on days 1, 2 and 3, IV.

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of benmelstobart in combination with anlotinib and chemotherapy sequential benmelstobart in combination with anlotinib for the first-line treatment of extensive-stage small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with pathologically confirmed extensive stage small cell lung cancer (VALG stage).
* 2. No prior systemic therapy for extensive-stage small cell lung cancer;
* 3. Patients who have received prior radiotherapy for limited-stage SCLC must have received radical therapy with a treatment-free interval of at least 6 months between the end of chemotherapy, radiotherapy, or radiochemotherapy and the diagnosis of extensive-stage SCLC (counting the time of completion of the last cycle of chemotherapy/time of completion of the last dose of radiotherapy);
* 4. The presence of a Measurable lesions as defined by the RECIST 1.1 criteria, where a previously irradiated lesion shows definite progression after radiotherapy and where this previously irradiated lesion is not the only lesion;
* 5. 18-75 years of age or older; ECOG score: 0-1; expected survival ≥ 3 months.
* 6. Adequate hematology and organ function, i.e., the following criteria are met:

  a) Hematology (no transfusion of blood or blood products within 14 days, not corrected with G-CSF and other hematopoietic stimulating factors): i. Absolute neutrophil count (ANC) ≥ 1.5 × 109/L (1,500/mm3); ii. Platelet count (PLT) ≥ 100 × 109/L (100,000 /mm3); iii. Hemoglobin (HB) ≥ 80 g/L.

  b) Renal: i. Creatinine clearance* (CrCl) calculated ≥ 50 mL/min; ii. Urine Protein < 2+ or 24 hour (h) urine protein quantification < 1.0 g.

  c) Liver: i. Serum total bilirubin (TBil) ≤ 1.5 × ULN; ii. AST and ALT ≤ 2.5 × ULN; iii. serum albumin (ALB) ≥ 28 g/L.

  d) Coagulation: i. International Normalized Ratio (INR) and Activated Partial Thromboplastin Time (APTT) ≤ 1.5 × ULN.

  e) Cardiac Function: i. Left Ventricular Ejection Fraction (LVEF) ≥ 50%.
* 7, Subjects voluntarily enrolled in this study and signed an informed consent form, complied well and cooperated with the follow-up.

Exclusion Criteria:

* 1, Patients with symptomatic brain metastases. Brain metastatic lesions that have been treated and kept in a clinically stable state of symptoms for at least 1 month, and do not use steroids and anticonvulsant drugs for at least 1 month prior to entering the study can be enrolled;
* 2. Previous use of anti-angiogenic drugs such as anlotinib, apatinib, bevacizumab, or related immunotherapeutic drugs targeting PD-1, PD-L1, etc.;
* 3. Those who have a wide range of factors affecting oral administration of the medication (e.g., the inability to swallow, After gastrointestinal resection, chronic diarrhea and intestinal obstruction, etc.);
* 4. Uncontrollable pleural effusion, pericardial effusion, or ascites that requires repeated drainage;
* 5. Patients with imaging evidence of tumor invasion of important perivascular vessels, or patients who, in the judgment of the investigator, are at high risk of fatal hemorrhage due to tumor invasion of an important blood vessel during the follow-up period of the study;
* 6. Patients with a history of severe hemorrhagic tendency or coagulation dysfunction including, but not limited to, clinical symptoms within 3 months prior to entry into the study. Clinically significant hemoptysis (greater than one tablespoon of hemoptysis per day) within 3 months prior to enrollment; or clinically significant bleeding symptoms or bleeding tendency within 4 weeks prior to enrollment, such as peptic hemorrhage, hemorrhagic gastric ulcers (including gastrointestinal perforation and/or fistulae, except that gastrointestinal perforation or fistulae that have been surgically resected may be permitted to be enrolled), non-healing wounds, ulcers, or bone fracture;
* 7. Patients who have received major Surgical treatment, incisional biopsy, or significant traumatic injury within 28 days prior to enrollment;
* 8. Arterial/venous thrombotic events, such as cerebrovascular accidents (including transient ischemic attacks), deep vein thrombosis, and pulmonary embolism, within 6 months prior to enrollment;
* 9. Active autoimmune disease requiring systemic therapy (e.g., palliative medications, corticosteroids, or immunosuppressants) within 2 years of the first dose;
* 10. Increased risk associated with participation in the study or study drug; and Other conditions that increase the risk associated with participation in the study or the study drug and, in the investigator's judgment, make the patient unsuitable for enrollment in the study;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Approximately 7 months from treatment.
  The time from treatment to the first documented progressive disease (PD) assessed by the investigator according to RECIST 1.1 or death for any reason. Evaluated every 2 cycles/6 weeks on treatment and every 3 months in follow-up.

SECONDARY OUTCOMES:
Overall Survival (OS) | Approximately 14 months from treatment.
  The time from treatment to death due to any cause. Follow-up visits were made every 3 months after the end of treatment.
Objective Response Rate (ORR) | Approximately 12 weeks after the last participant begin study treatment.
  Percentage of participants who achieved Complete Response (CR) or Partial Response (PR), assessed by the investigator according to RECIST 1.1.
Duration of Response (DOR) | Approximately 7 months from treatment.
  The time from the first response (Complete Response (CR) or Partial Response (PR)) to disease progression (PD) assessed by the investigator according to RECIST 1.1 or death for any reason.
Disease Control Rate (DCR) | Approximately 12 weeks after the last participant begin study treatment.
  Percentage of participants who achieved Complete Response (CR), Partial Response (PR) or Stable Disease (SD), assessed by the investigator according to RECIST 1.1.
Safety (Adverse Events (AEs)) | From enrollment until 30 days after the end of treatment.
  Type and severity of adverse events according to CTCAE v5.0; calculation of the incidence of adverse events and their incidence by system.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided